CLINICAL TRIAL: NCT02024386
Title: The Effect of Riociguat on Gas Exchange, Exercise Performance, and Pulmonary Artery Pressure During Acute Altitude Exposure
Brief Title: Efficacy Study of Riociguat and Its Effects on Exercise Performance and Pulmonary Artery Pressure at High Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Moon (Other)
Responsible Party: Sponsor-Investigator, Richard Moon, Medical Director, Duke Center for Hyperbaric Medicine and Environmental Physiology, Professor of Anesthesiology, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00049150
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Hypertension, Pulmonary; Altitude Sickness
Keywords: Guanylate Cyclase; Pulmonary Edema of Mountaineers; Mountaineering; Performance-Enhancing Substances; Athletic Performance
MeSH Terms: conditions — Hypertension, Pulmonary; Altitude Sickness; Pulmonary edema of mountaineers | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Riociguat 0.5 mg (Experimental): Riociguat 0.5 mg tablets, one-time oral dose of 0.5 mg
  Interventions: Drug: Riociguat
- Riociguat 1.0 mg (Experimental): Riociguat 0.5 mg tablets, one-time oral dose of 1.0 mg
  Interventions: Drug: Riociguat
- Control arm (No Intervention): No drug

INTERVENTIONS:
Drug: Riociguat — After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. Riociguat will be administered at the 90-minute mark of this rest period.
  Other Names: Adempas; NDA 204819
  Arms: Riociguat 0.5 mg; Riociguat 1.0 mg

SUMMARY:
During ascent to high altitude there is a physiologic response to hypoxia that results in an elevated pulmonary arterial pressure associated with decreased exercise performance, altitude-induced pulmonary hypertension, and high altitude pulmonary edema (HAPE). Riociguat is a novel agent from Bayer Pharmaceuticals that has already demonstrated effectiveness in the treatment of pulmonary hypertension, and it may prove to be beneficial in cases of altitude-induced pulmonary hypertension or HAPE. This research study, composed of 20 healthy volunteers ages 18-40 years, will attempt to mimic the decreased oxygen supply and elevated pulmonary artery pressures found in conditions of high altitude, allowing observation of the effects of riociguat and exercise on pulmonary arterial pressure, arterial oxygenation, and exercise performance. Prior to entering the hypobaric chamber, subjects will have radial arterial lines and pulmonary artery catheters placed to obtain arterial and pulmonary artery pressure measurements. Subjects will then enter the hypobaric chamber and perform exercise tolerance tests at a simulated altitude of 15,000 feet on an electrically braked ergometer (exercise bike) before and after administration of riociguat. If, after administration of riociguat and exposure to a simulated altitude of 15,000 feet, the exercise performance is improved and observed pulmonary artery pressures are lower than those measurements seen prior to administration of riociguat, this could lead to development of a prophylactic and/or treatment strategy for HAPE and high-altitude pulmonary hypertension. Statistical analysis will compare the variables of pulmonary artery pressure, radial arterial pressure, ventilation rate, cardiac output, PaO2, and work rate at exhaustion before and after administration of the drug riociguat. The investigator's hypothesis is that riociguat will decrease pulmonary artery pressure and improve gas exchange and exercise performance at altitude.

DETAILED DESCRIPTION:
Background and Significance:

Impairment of exercise performance during hypoxemia due to altitude exposure or lung disease is caused primarily by reduced oxygen delivery to the exercising muscles, due to the reduction in arterial oxygen content. This reduction in arterial oxygen content is due to reduced alveolar PO2 and ventilation/perfusion (VA/Q) mismatch, and to some extent alveolar to end-capillary diffusion impairment. Ultimately, hypoxemia results in secondary diffuse pulmonary vasoconstriction (hypoxic pulmonary vasoconstriction, HPV), which in turn causes pulmonary hypertension. This secondary pulmonary hypertension is believed to worsen VA/Q mismatch, further reducing the PO2, suggesting that pharmacologic blockade of HPV could increase PO2 (e.g. during altitude exposure) and thus improve exercise performance. Reduction in pulmonary artery pressure (PAP) in individuals susceptible to high altitude pulmonary edema (HAPE) could also facilitate both prevention and treatment of HAPE.

Sildenafil is commonly used to treat pulmonary hypertension, including pulmonary hypertension that occurs due to altitude exposure, with variable success in treating cases of altitude-induced pulmonary hypertension and HAPE. Sildenafil works via blockade of blocks phosphodiesterase-5 (PDE-5) in pulmonary arterioles, causing an increase in cGMP. When cGMP is activated by nitric oxide (NO) it induces vasodilatation, and indeed, sildenafil administration during altitude exposure does increase arterial oxygenation slightly. However, attempting to block HPV with sildenafil by using a pathway that requires NO can only be realized if there is sufficient NO available to produce cGMP. During hypoxia endogenous levels of NO are depleted due to impaired endothelial NO synthesis. This may explain the inconsistent effects of sildenafil when used to improve oxygenation and performance at altitude.

Endogenous concentration of unbound NO is actually quite low, and most of the biological effects of NO are mediated through formation of S-nitrosothiols (SNOs) such as S-nitrosohemoglobin (SNO-Hb). NO binds to hemoglobin in a PO2-dependent manner, forming SNO-Hb so that when PO2 is low, NO-Hb binding is less avid and SNO-Hb is depleted. Depletion of SNO-Hb during hypoxia has been proposed as a mechanism that augments HPV, and indeed hypoxia has been shown to induce low levels of SNO-Hb. It is quite possible that the reduction in available endogenous NO and depletion of SNO-Hb during hypoxia limits the effect of the cGMP mechanism by which sildenafil works. Thus, an agent which can activate cGMP during periods of hypoxia when NO and SNO-Hb are depleted should be more effective in treating altitude-induced pulmonary hypertension.

Riociguat is a stimulator of soluble guanylate cyclase that bypasses the NO pathway and is currently approved by the FDA for treatment of pulmonary hypertension. Riociguat exhibits a dual mode of action that i.) stabilizes the reduced form of the nitrosyl-heme complex, enhancing the NO-cGMP signaling pathway in the absence of endogenous NO and ii.) acts in synergy with endogenous NO by increasing sGC sensitivity to NO. Essentially, riociguat stimulates sGC to produce cGMP in the absence of NO, and it is a mechanism by which pulmonary vascular resistance could be attenuated during altitude-induced pulmonary hypertension. It has recently been shown to augment exercise performance and decrease pulmonary artery pressure in both primary pulmonary hypertension and pulmonary arterial hypertension (PAH) due to chronic thromboembolic disease. Lowering pulmonary artery pressure could improve pulmonary gas exchange and performance at altitude, which has significant implications for those living at altitude, conducting military operations, altitude trekkers and high-altitude rescue teams. Direct stimulation of sGC also represents a promising alternative therapeutic strategy for those susceptible to high altitude pulmonary edema (HAPE) when current treatment modalities of nifedipine and sildenafil are ineffective and oxygen is unavailable. By itself or in combination with sildenafil, riociguat could produce a significant advance in exercise performance during altitude exposure and provide a substantial improvement over the current therapeutic options in the prevention and treatment of HAPE.

Design and Procedures:

This investigation will consist of 20 normal subjects. Medical screening will exclude cardiac and pulmonary disease, pregnancy and sickle cell disease/trait in African Americans.

Subjects will be instrumented with radial arterial lines and pulmonary artery catheters and will perform a VO2 max test on a bicycle ergometer in a hypobaric chamber at a simulated altitude of 15,000 feet.

Following the VO2 max test, subjects will return to ground level for a 3-hour rest period. At 90 minutes subjects will be administered riociguat 0.5 mg or 1.0 mg orally. Once study subjects are at therapeutic levels of riociguat (30 to 90 minutes after oral administration), they will repeat the VO2 max test at 15,000 feet. The dosing of riociguat will start at the lowest recommended individual dose (0.5 mg) for the first three subjects. If there are no side effects and no clinically important difference in either PAP (5 mmHg decrease in mean PAP) or PaO2 (5 mmHg increase) during exercise, then for the remaining subjects the dose will be increased to 1.0 mg.

During the incremental exercise test arterial and mixed blood samples will be analyzed for PO2, PCO2, pH, O2 saturation and hemoglobin. Exhaled gas will be collected continuously and analyzed for O2 and CO2 concentrations and exhaled volume. Cardiac output will be calculated using Fick. Pulmonary and systemic vascular resistances will be calculated from the cardiac output and intravascular pressures.

Outcome measures will be VO2max, maximum mechanical work rate, pulmonary and systemic arterial pressures, cardiac output, oxygen delivery and arterial blood gases.

Benefits:

Further understanding of the mechanism of hypoxic pulmonary vasoconstriction will aid in prognosis and treatment in conditions of increased pulmonary vascular resistance such as congenital heart disease, pulmonary arterial hypertension, and COPD, in addition to high-altitude pulmonary hypertension and high-altitude pulmonary edema (HAPE). Furthermore, the current treatment modalities for HAPE have demonstrated variable and/or limited effectiveness, so riociguat could potentially be used to prevent or treat HAPE in susceptible individuals. Additionally, riociguat could substantially improve exercise performance in those who must operate in conditions of high-altitude, such as those conducting military operations or working in high-altitude rescue teams.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Non-smoking
* Non-pregnant females
* Ages 18 - 40 years old

Exclusion Criteria:

* Serious pulmonary or cardiovascular comorbidities
* Pregnant women
* VO2max < 35 mL/kg per minute
* Sickle cell trait or disease
* Smokers
* Lung disease
* Hypertension
* Cardiac disease and left bundle branch block
* Taking nitrates, nitric oxide donors (such as amyl nitrite), and phosphodiesterase (PDE) inhibitors (including specific PDE-5 inhibitors, such as sildenafil, tadalafil, or vardenafil, or non-specific PDE inhibitors, such as dipyridamole or theophylline).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Moon, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Hyperbaric Medicine and Environmental Physiology, Trent Drive, Building CR2, Room 0584, Box 3823,, Durham, North Carolina, United States

REFERENCES:
- [Background] Torre-Bueno JR, Wagner PD, Saltzman HA, Gale GE, Moon RE. Diffusion limitation in normal humans during exercise at sea level and simulated altitude. J Appl Physiol (1985). 1985 Mar;58(3):989-95. doi: 10.1152/jappl.1985.58.3.989. PMID 2984169
- [Background] Gale GE, Torre-Bueno JR, Moon RE, Saltzman HA, Wagner PD. Ventilation-perfusion inequality in normal humans during exercise at sea level and simulated altitude. J Appl Physiol (1985). 1985 Mar;58(3):978-88. doi: 10.1152/jappl.1985.58.3.978. PMID 2984168
- [Background] Wagner PD, Gale GE, Moon RE, Torre-Bueno JR, Stolp BW, Saltzman HA. Pulmonary gas exchange in humans exercising at sea level and simulated altitude. J Appl Physiol (1985). 1986 Jul;61(1):260-70. doi: 10.1152/jappl.1986.61.1.260. PMID 3090012
- [Background] Ghofrani HA, Reichenberger F, Kohstall MG, Mrosek EH, Seeger T, Olschewski H, Seeger W, Grimminger F. Sildenafil increased exercise capacity during hypoxia at low altitudes and at Mount Everest base camp: a randomized, double-blind, placebo-controlled crossover trial. Ann Intern Med. 2004 Aug 3;141(3):169-77. doi: 10.7326/0003-4819-141-3-200408030-00005. PMID 15289213
- [Background] Richalet JP, Gratadour P, Robach P, Pham I, Dechaux M, Joncquiert-Latarjet A, Mollard P, Brugniaux J, Cornolo J. Sildenafil inhibits altitude-induced hypoxemia and pulmonary hypertension. Am J Respir Crit Care Med. 2005 Feb 1;171(3):275-81. doi: 10.1164/rccm.200406-804OC. Epub 2004 Oct 29. PMID 15516532
- [Background] McMahon TJ, Moon RE, Luschinger BP, Carraway MS, Stone AE, Stolp BW, Gow AJ, Pawloski JR, Watke P, Singel DJ, Piantadosi CA, Stamler JS. Nitric oxide in the human respiratory cycle. Nat Med. 2002 Jul;8(7):711-7. doi: 10.1038/nm718. Epub 2002 Jun 3. PMID 12042776
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] McMahon TJ, Ahearn GS, Moya MP, Gow AJ, Huang YC, Luchsinger BP, Nudelman R, Yan Y, Krichman AD, Bashore TM, Califf RM, Singel DJ, Piantadosi CA, Tapson VF, Stamler JS. A nitric oxide processing defect of red blood cells created by hypoxia: deficiency of S-nitrosohemoglobin in pulmonary hypertension. Proc Natl Acad Sci U S A. 2005 Oct 11;102(41):14801-6. doi: 10.1073/pnas.0506957102. Epub 2005 Oct 3. PMID 16203976
- [Background] Allen BW, Stamler JS, Piantadosi CA. Hemoglobin, nitric oxide and molecular mechanisms of hypoxic vasodilation. Trends Mol Med. 2009 Oct;15(10):452-60. doi: 10.1016/j.molmed.2009.08.002. Epub 2009 Sep 24. PMID 19781996
- [Background] Rubin LJ, Naeije R. Sildenafil for enhanced performance at high altitude? Ann Intern Med. 2004 Aug 3;141(3):233-5. doi: 10.7326/0003-4819-141-3-200408030-00016. No abstract available. PMID 15289224
- [Background] Droma Y, Hanaoka M, Ota M, Katsuyama Y, Koizumi T, Fujimoto K, Kobayashi T, Kubo K. Positive association of the endothelial nitric oxide synthase gene polymorphisms with high-altitude pulmonary edema. Circulation. 2002 Aug 13;106(7):826-30. doi: 10.1161/01.cir.0000024409.30143.70. PMID 12176955
- [Background] Ahsan A, Charu R, Pasha MA, Norboo T, Charu R, Afrin F, Ahsan A, Baig MA. eNOS allelic variants at the same locus associate with HAPE and adaptation. Thorax. 2004 Nov;59(11):1000-2. doi: 10.1136/thx.2004.029124. No abstract available. PMID 15516480
- [Background] Luo Y, Chen Y, Zhang Y, Zhou Q, Gao Y. Association of endothelial nitric oxide synthase (eNOS) G894T polymorphism with high altitude pulmonary edema susceptibility: a meta-analysis. Wilderness Environ Med. 2012 Sep;23(3):270-4. doi: 10.1016/j.wem.2012.03.007. Epub 2012 Jul 13. PMID 22795910
- [Background] Follmann M, Griebenow N, Hahn MG, Hartung I, Mais FJ, Mittendorf J, Schafer M, Schirok H, Stasch JP, Stoll F, Straub A. The chemistry and biology of soluble guanylate cyclase stimulators and activators. Angew Chem Int Ed Engl. 2013 Sep 2;52(36):9442-62. doi: 10.1002/anie.201302588. Epub 2013 Aug 20. PMID 23963798
- [Background] Ghofrani HA, D'Armini AM, Grimminger F, Hoeper MM, Jansa P, Kim NH, Mayer E, Simonneau G, Wilkins MR, Fritsch A, Neuser D, Weimann G, Wang C; CHEST-1 Study Group. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension. N Engl J Med. 2013 Jul 25;369(4):319-29. doi: 10.1056/NEJMoa1209657. PMID 23883377
- [Background] Ghofrani HA, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh AM, Langleben D, Kilama MO, Fritsch A, Neuser D, Rubin LJ; PATENT-1 Study Group. Riociguat for the treatment of pulmonary arterial hypertension. N Engl J Med. 2013 Jul 25;369(4):330-40. doi: 10.1056/NEJMoa1209655. PMID 23883378
- [Background] Forster PJ. Effect of different ascent profiles on performance at 4,200 m elevation. Aviat Space Environ Med. 1985 Aug;56(8):758-64. PMID 3929759
- [Background] West JB. Improving oxygenation at high altitude: acclimatization and O2 enrichment. High Alt Med Biol. 2003 Fall;4(3):389-98. doi: 10.1089/152702903769192340. PMID 14561244
- [Background] Beidleman BA, Muza SR, Fulco CS, Cymerman A, Ditzler D, Stulz D, Staab JE, Skrinar GS, Lewis SF, Sawka MN. Intermittent altitude exposures reduce acute mountain sickness at 4300 m. Clin Sci (Lond). 2004 Mar;106(3):321-8. doi: 10.1042/CS20030161. PMID 14561214
- [Background] Sampson JB, Cymerman A, Burse RL, Maher JT, Rock PB. Procedures for the measurement of acute mountain sickness. Aviat Space Environ Med. 1983 Dec;54(12 Pt 1):1063-73. PMID 6661120
- [Background] Rock PB, Johnson TS, Cymerman A, Burse RL, Falk LJ, Fulco CS. Effect of dexamethasone on symptoms of acute mountain sickness at Pikes Peak, Colorado (4,300 m). Aviat Space Environ Med. 1987 Jul;58(7):668-72. PMID 3619842
- [Background] Hughson RL, Yamamoto Y, McCullough RE, Sutton JR, Reeves JT. Sympathetic and parasympathetic indicators of heart rate control at altitude studied by spectral analysis. J Appl Physiol (1985). 1994 Dec;77(6):2537-42. doi: 10.1152/jappl.1994.77.6.2537. PMID 7896588
- [Background] Bartsch P, Maggiorini M, Ritter M, Noti C, Vock P, Oelz O. Prevention of high-altitude pulmonary edema by nifedipine. N Engl J Med. 1991 Oct 31;325(18):1284-9. doi: 10.1056/NEJM199110313251805. PMID 1922223
- [Background] Scherrer U, Vollenweider L, Delabays A, Savcic M, Eichenberger U, Kleger GR, Fikrle A, Ballmer PE, Nicod P, Bartsch P. Inhaled nitric oxide for high-altitude pulmonary edema. N Engl J Med. 1996 Mar 7;334(10):624-9. doi: 10.1056/NEJM199603073341003. PMID 8592525
- [Background] Jensen LA, Onyskiw JE, Prasad NG. Meta-analysis of arterial oxygen saturation monitoring by pulse oximetry in adults. Heart Lung. 1998 Nov-Dec;27(6):387-408. doi: 10.1016/s0147-9563(98)90086-3. PMID 9835670
- [Background] Hornbein TF, Townes BD, Schoene RB, Sutton JR, Houston CS. The cost to the central nervous system of climbing to extremely high altitude. N Engl J Med. 1989 Dec 21;321(25):1714-9. doi: 10.1056/NEJM198912213212505. PMID 2512483
- [Background] Frey R, Muck W, Unger S, Artmeier-Brandt U, Weimann G, Wensing G. Single-dose pharmacokinetics, pharmacodynamics, tolerability, and safety of the soluble guanylate cyclase stimulator BAY 63-2521: an ascending-dose study in healthy male volunteers. J Clin Pharmacol. 2008 Aug;48(8):926-34. doi: 10.1177/0091270008319793. Epub 2008 Jun 2. PMID 18519919
- [Background] Slogoff S, Keats AS, Arlund C. On the safety of radial artery cannulation. Anesthesiology. 1983 Jul;59(1):42-7. doi: 10.1097/00000542-198307000-00008. PMID 6859611
- [Background] Frezza EE, Mezghebe H. Indications and complications of arterial catheter use in surgical or medical intensive care units: analysis of 4932 patients. Am Surg. 1998 Feb;64(2):127-31. PMID 9486883
- [Background] Valentine RJ, Modrall JG, Clagett GP. Hand ischemia after radial artery cannulation. J Am Coll Surg. 2005 Jul;201(1):18-22. doi: 10.1016/j.jamcollsurg.2005.01.011. PMID 15978439
- [Background] Mummery HJ, Stolp BW, deL Dear G, Doar PO, Natoli MJ, Boso AE, Archibald JD, Hobbs GW, El-Moalem HE, Moon RE. Effects of age and exercise on physiological dead space during simulated dives at 2.8 ATA. J Appl Physiol (1985). 2003 Feb;94(2):507-17. doi: 10.1152/japplphysiol.00367.2002. Epub 2002 Oct 11. PMID 12391136

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six additional subjects were consented but not enrolled. Two subjects failed the screen due to a VO2 max less than the inclusion criteria. Two subjects were withdrawn when the Swan-Ganz catheter could not be placed. One subject was unable to schedule an experimental date and one subject did not return for screening.
Groups:
- Riociguat 0.5 mg: Riociguat 0.5 mg tablets, one-time oral dose of 0.5
  Riociguat: After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. A second VO2 max test will be repeated at altitude 90 minutes after Riociguat administration.
- Riociguat 1.0 mg: Riociguat 0.5 mg tablets, one-time oral dose of 1.0 mg
  Riociguat: After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. A second VO2 max test will be repeated at altitude 90 minutes after Riociguat administration.
- Control Arm: No drug
  After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. A second VO2 max test will be repeated at altitude.
Period: Overall Study
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Started | 6 | 11 | 5
Completed | 6 | 11 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm | Total
Number analyzed (Participants) | 6 | 11 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.2) | 24.3 (4.4) | 24.8 (5.2) | 26.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 4
  Male | 6 | 7 | 5 | 18
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Pulmonary Artery Pressure
Description: Subject pulmonary artery pressures will be continuously monitored during the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Exercise level will be increased every 3 minutes until test termination criteria are achieved. Measurements will be obtained at rest, every 3 minutes during the exercise test (referred to as a stage below) and at 5 minutes post exercise. Results will be reported as a 30 second average. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
mm Hg
  No Drug: Rest | 16.8667 (4.82604) | 15.6545 (4.93728) | 16.3800 (3.11400)
  After Drug: Rest: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Rest | 16.6833 (1.41622) | 15.4900 (5.14078) | 17.4000 (3.57980)
  No Drug: Stage 1 | 25.0000 (3.93904) | 26.9455 (7.21074) | 25.3600 (5.10225)
  After Drug: Stage 1 | 26.1167 (3.09866) | 25.1545 (6.54437) | 25.0800 (5.02215)
  No Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  No Drug: Stage 2 | 27.2800 (2.66402) | 26.5800 (4.53696) | 26.6600 (4.19321)
  After Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  After Drug: Stage 2 | 27.0600 (2.38181) | 25.5100 (4.41121) | 27.4400 (4.26063)
  No Drug: Stage 3: number analyzed (Participants) | 5 | 9 | 4
  No Drug: Stage 3 | 28.0200 (2.09929) | 26.4111 (3.68627) | 25.7000 (1.61038)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 4
  After Drug: Stage 3 | 28.0500 (2.59037) | 24.1375 (3.13184) | 26.8500 (3.60509)
  No Drug: Stage 4: number analyzed (Participants) | 5 | 8 | 4
  No Drug: Stage 4 | 29.7400 (3.19421) | 27.2750 (3.72702) | 26.9750 (1.32004)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 4
  After Drug: Stage 4 | 29.3750 (2.38939) | 25.2167 (3.90662) | 27.4000 (4.27785)
  No Drug: Stage 5: number analyzed (Participants) | 5 | 11 | 4
  No Drug: Stage 5 | 30.8400 (2.67638) | 28.0333 (4.54914) | 27.5000 (0.87560)
  After Drug: Stage 5: number analyzed (Participants) | 2 | 5 | 4
  After Drug: Stage 5 | 28.5000 (0.42426) | 24.2000 (3.57561) | 28.1500 (3.63089)
  No Drug: Stage 6: number analyzed (Participants) | 4 | 4 | 3
  No Drug: Stage 6 | 32.6500 (3.59119) | 25.9250 (3.73932) | 28.7667 (2.00083)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 36.1000 (0) | 22.7000 (4.82563) | 29.4333 (3.25167)
  No Drug: Stage 7: number analyzed (Participants) | 3 | 2 | 1
  No Drug: Stage 7 | 32.9333 (3.62537) | 20.4000 (0.98995) | 26.6000
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 22.5000 (4.38406) |
  No Drug: Post Exercise: number analyzed (Participants) | 6 | 10 | 5
  No Drug: Post Exercise | 18.9500 (1.49766) | 19.1273 (3.54375) | 19.3000 (3.41541)
  After Drug: Post Exercise: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Post Exercise | 19.2167 (3.20962) | 16.6700 (3.53303) | 19.2800 (3.98083)

2. Secondary Outcome: Mean Radial Arterial Pressure
Description: Subject systemic arterial pressures will be continuously monitored via radial artery catheterization during the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Exercise level will be increased every 3 minutes until test termination criteria are achieved. Measurements will be obtained at rest, every 3 minutes during the exercise test (referred to as a stage below) and at 5 minutes post exercise. Results will be reported as a 30 second average. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
mm Hg
  No Drug: Rest | 87.8333 (7.50697) | 93.3182 (6.88474) | 96.5600 (3.94310)
  After Drug: Rest: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Rest | 91.6000 (6.68820) | 91.8000 (7.96171) | 96.7600 (7.87102)
  No Drug: Stage 1 | 93.5167 (9.2227) | 101.545 (6.19231) | 100.1600 (12.2541)
  After Drug: Stage 1 | 97.1167 (11.6199) | 97.627 (7.23645) | 102.500 (13.6998)
  No Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  No Drug: Stage 2 | 105.480 (7.23063) | 107.270 (4.49074) | 107.020 (12.4432)
  After Drug: Stage 2: number analyzed (Participants) | 5 | 9 | 5
  After Drug: Stage 2 | 107.260 (8.15494) | 104.867 (4.38834) | 105.580 (16.6067)
  No Drug: Stage 3: number analyzed (Participants) | 5 | 9 | 4
  No Drug: Stage 3 | 107.580 (7.0733) | 110.122 (6.10794) | 109.425 (14.9402)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 4
  After Drug: Stage 3 | 114.65 (10.2142) | 106.425 (6.00541) | 111.825 (17.3803)
  No Drug: Stage 4: number analyzed (Participants) | 5 | 8 | 4
  No Drug: Stage 4 | 113.140 (7.43962) | 114.650 (6.39710) | 112.675 (13.6754)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 4
  After Drug: Stage 4 | 117.025 (9.37386) | 109.517 (8.24874) | 112.475 (18.1522)
  No Drug: Stage 5: number analyzed (Participants) | 5 | 6 | 4
  No Drug: Stage 5 | 116.500 (9.67471) | 115.267 (9.39184) | 114.775 (12.2004)
  After Drug: Stage 5: number analyzed (Participants) | 2 | 5 | 4
  After Drug: Stage 5 | 124.800 (8.76812) | 108.240 (9.10950) | 114.175 (14.4756)
  No Drug: Stage 6: number analyzed (Participants) | 4 | 4 | 3
  No Drug: Stage 6 | 115.900 (13.4291) | 112.025 (9.61852) | 108.100 (3.89744)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 143.1 | 108.825 (9.33323) | 107.367 (5.40031)
  No Drug: Stage 7: number analyzed (Participants) | 3 | 2 | 1
  No Drug: Stage 7 | 122.700 (21.3551) | 107.900 (5.23259) | 101.9
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 102.400 (7.91960) |
  No Drug: Post Exercise | 89.500 (9.01665) | 90.3545 (15.1484) | 90.4800 (17.2794)
  After Drug: Post Exercise: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Post Exercise | 92.0833 (5.13358) | 81.7800 (12.2102) | 95.3600 (13.4986)

3. Secondary Outcome: Mean Arterial Oxygen Saturation (SaO2)
Description: Subject arterial oxygen saturation (SaO2) will be periodically monitored at fixed intervals via arterial blood gas measurements during the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Measurements will be obtained at rest, every 3 minutes during the exercise test (referred to as a stage below) and at 5 minutes post exercise. Results will be reported as a 30 second average. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: % oxygen saturation
Groups:
- Riociguat 0.5 mg: Riociguat 0.5 mg tablets, one-time oral dose of 0.5 mg
  Riociguat: After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. A second VO2 max test will be repeated at altitude 90 minutes after Riociguat administration.
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
% oxygen saturation
  No Drug: Rest | 78.3333 (5.73957) | 84.9364 (6.87696) | 85.4400 (6.50215)
  After Drug: Rest: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Rest | 81.9667 (6.93186) | 84.4000 (6.56624) | 83.9000 (3.88909)
  No Drug: Stage 1: number analyzed (Participants) | 5 | 11 | 5
  No Drug: Stage 1 | 71.2800 (4.90683) | 73.1545 (7.01703) | 74.2600 (5.79552)
  After Drug: Stage 1: number analyzed (Participants) | 5 | 10 | 5
  After Drug: Stage 1 | 72.5800 (3.89460) | 74.0000 (7.14967) | 70.9800 (6.00267)
  No Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  No Drug: Stage 2 | 71.0800 (0.67971) | 72.4800 (7.56862) | 70.9200 (5.23612)
  After Drug: Stage 2: number analyzed (Participants) | 4 | 9 | 5
  After Drug: Stage 2 | 73.4500 (3.17753) | 74.2556 (7.88339) | 69.9800 (6.53506)
  No Drug: Stage 3: number analyzed (Participants) | 4 | 9 | 4
  No Drug: Stage 3 | 71.5250 (2.65503) | 71.9333 (7.44681) | 67.1750 (6.63193)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 4
  After Drug: Stage 3 | 72.2500 (3.79956) | 73.5000 (8.83823) | 67.7500 (7.50533)
  No Drug: Stage 4: number analyzed (Participants) | 5 | 8 | 4
  No Drug: Stage 4 | 71.3400 (2.39958) | 72.1250 (7.55735) | 68.9500 (8.11521)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 4
  After Drug: Stage 4 | 70.9000 (2.48956) | 72.0167 (8.17103) | 68.3500 (7.91686)
  No Drug: Stage 5: number analyzed (Participants) | 4 | 6 | 4
  No Drug: Stage 5 | 71.3250 (3.20975) | 69.6333 (6.37139) | 68.825 (8.07687)
  After Drug: Stage 5: number analyzed (Participants) | 2 | 5 | 4
  After Drug: Stage 5 | 70.1000 (0.84853) | 72.5200 (6.68731) | 68.825 (8.26131)
  No Drug: Stage 6: number analyzed (Participants) | 4 | 4 | 3
  No Drug: Stage 6 | 71.5000 (2.88560) | 71.4750 (3.61513) | 66.5000 (7.83071)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 67.3000 | 71.9750 (2.98035) | 64.8667 (6.24206)
  No Drug: Stage 7: number analyzed (Participants) | 3 | 2 | 1
  No Drug: Stage 7 | 73.9667 (7.80790) | 70.8500 (1.20208) | 67.7000
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 68.7000 (0.14142) |
  No Drug: Post Exercise | 76.3500 (6.30325) | 79.2182 (4.72479) | 82.0400 (4.10889)
  After Drug: Post Exercise: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Post Exercise | 80.5833 (5.78983) | 81.2700 (3.60341) | 83.5400 (5.50799)

4. Secondary Outcome: Mean Ventilation Rate
Description: Subject ventilation rates will be monitored continuously using a multi-channel A/D converter (PowerLab™) connected to a personal computer, using Chart™ software (ADInstruments, Colorado Springs, CO) during the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Exercise level will be increased every 3 minutes until test termination criteria are achieved. Measurements will be obtained at rest, every 3 minutes during the exercise test (referred to as a stage below) and at 5 minutes post exercise. Results will be reported as a 30 second average. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
L/min
  No Drug: Rest: number analyzed (Participants) | 5 | 11 | 5
  No Drug: Rest | 14.7634 (2.43930) | 16.8981 (5.52822) | 18.2266 (5.08350)
  After Drug: Rest: number analyzed (Participants) | 5 | 9 | 4
  After Drug: Rest | 17.5454 (3.71867) | 18.9289 (8.96658) | 16.4128 (4.11186)
  No Drug: Stage 1: number analyzed (Participants) | 5 | 11 | 5
  No Drug: Stage 1 | 38.3134 (8.3828) | 40.8095 (9.07931) | 46.0238 (5.20868)
  After Drug: Stage 1: number analyzed (Participants) | 6 | 11 | 4
  After Drug: Stage 1 | 40.3488 (12.2484) | 41.3605 (5.52287) | 42.0435 (7.34401)
  No Drug: Stage 2: number analyzed (Participants) | 4 | 10 | 5
  No Drug: Stage 2 | 52.1473 (3.73255) | 64.6476 (11.3309) | 63.2124 (14.8132)
  After Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 4
  After Drug: Stage 2 | 59.9588 (3.22699) | 61.4905 (10.9421) | 60.8040 (12.9110)
  No Drug: Stage 3: number analyzed (Participants) | 4 | 9 | 4
  No Drug: Stage 3 | 67.3315 (3.16166) | 81.5548 (11.9696) | 70.9060 (2.74032)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 3
  After Drug: Stage 3 | 73.6560 (8.62422) | 78.0649 (10.5961) | 69.1603 (5.38746)
  No Drug: Stage 4: number analyzed (Participants) | 4 | 8 | 4
  No Drug: Stage 4 | 89.7233 (8.06763) | 102.499 (13.8660) | 89.3008 (5.95060)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 3
  After Drug: Stage 4 | 97.2645 (9.83327) | 96.850 (10.1315) | 92.8173 (7.48757)
  No Drug: Stage 5: number analyzed (Participants) | 4 | 6 | 4
  No Drug: Stage 5 | 108.857 (9.0793) | 132.789 (19.6447) | 113.354 (9.9434)
  After Drug: Stage 5: number analyzed (Participants) | 3 | 5 | 3
  After Drug: Stage 5 | 121.556 (25.4212) | 126.372 (11.5500) | 118.521 (16.2642)
  No Drug: Stage 6: number analyzed (Participants) | 3 | 4 | 3
  No Drug: Stage 6 | 143.373 (7.76136) | 153.233 (19.5104) | 137.837 (19.5282)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 145.65 | 151.843 (21.1490) | 134.869 (10.3445)
  No Drug: Stage 7: number analyzed (Participants) | 2 | 2 | 1
  No Drug: Stage 7 | 156.669 (14.2390) | 173.819 (20.2664) | 126.447
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 156.978 (7.9330) |
  No Drug: Post Exercise: number analyzed (Participants) | 3 | 10 | 5
  No Drug: Post Exercise | 32.3927 (7.0137) | 38.1639 (20.6608) | 41.7934 (10.1981)
  After Drug: Post Exercise: number analyzed (Participants) | 5 | 9 | 4
  After Drug: Post Exercise | 29.6728 (11.2070) | 34.7268 (13.9398) | 40.7953 (6.8369)

5. Secondary Outcome: Mean Work Rate at Exhaustion
Description: Subject work rates at exhaustion (in watts) will be continuously monitored using an ergometer (exercise bicycle) during the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Exercise level will be increased every 3 minutes until test termination criteria are achieved. Measurements will be obtained at rest, every 3 minutes during the exercise test (referred to as a stage below) and at 5 minutes post exercise. Results will be reported as a 30 second average. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
watts
  No Drug: Rest | 0 (0) | 0 (0) | 0 (0)
  After Drug: Rest | 0 (0) | 0 (0) | 0 (0)
  No Drug: Stage 1 | 50 (0) | 50 (0) | 50 (0)
  After Drug: Stage 1: number analyzed (Participants) | 6 | 10 | 5
  After Drug: Stage 1 | 50 (0) | 50 (0) | 50 (0)
  No Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  No Drug: Stage 2 | 75 (0) | 75 (0) | 75 (0)
  After Drug: Stage 2: number analyzed (Participants) | 5 | 10 | 5
  After Drug: Stage 2 | 75 (0) | 75 (0) | 75 (0)
  No Drug: Stage 3: number analyzed (Participants) | 5 | 9 | 4
  No Drug: Stage 3 | 100 (0) | 100 (0) | 100 (0)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 4
  After Drug: Stage 3 | 100 (0) | 100 (0) | 100 (0)
  No Drug: Stage 4: number analyzed (Participants) | 5 | 8 | 4
  No Drug: Stage 4 | 125 (0) | 125 (0) | 125 (0)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 4
  After Drug: Stage 4 | 125 (0) | 125 (0) | 125 (0)
  No Drug: Stage 5: number analyzed (Participants) | 5 | 6 | 4
  No Drug: Stage 5 | 150 (0) | 150 (0) | 150 (0)
  After Drug: Stage 5: number analyzed (Participants) | 3 | 5 | 4
  After Drug: Stage 5 | 150 (0) | 150 (0) | 150 (0)
  No Drug: Stage 6: number analyzed (Participants) | 4 | 4 | 3
  No Drug: Stage 6 | 175 (0) | 175 (0) | 175 (0)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 175 (0) | 175 (0) | 175 (0)
  No Drug: Stage 7: number analyzed (Participants) | 3 | 2 | 1
  No Drug: Stage 7 | 200 (0) | 200 (0) | 200 (0)
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 200 (0) |
  No Drug: Post Exercise: number analyzed (Participants) | 5 | 11 | 4
  No Drug: Post Exercise | 0 (0) | 0 (0) | 0 (0)
  After Drug: Post Exercise: number analyzed (Participants) | 6 | 9 | 5
  After Drug: Post Exercise | 0 (0) | 0 (0) | 0 (0)

6. Secondary Outcome: Cardiac Output
Description: Arterial blood samples will be obtained before, during, and after the VO2max exercise test in the hypobaric chamber at a simulated altitude of 15,000 feet. Exercise level will be increased every 3 minutes until test termination criteria are achieved. Samples will be obtained during the fifth minute of rest prior to exercise, during the third minute of each exercise level (referred to as stage below) and during the fifth minute post exercise. Cardiac output (CO) will be calculated using the Fick Principle: CO = V̇O2/(CaO2 - Cv̄O2) where CaO2 and Cv̄O2 represent the arterial and mixed venous oxygen content, respectively. CaO2 and CvO2 will be determined from analysis of the arterial blood samples using an IL GEM 4000 analyzer. VO2 will be reported as the final 30 secon average value of each stage. Subjects in the Riociguat cohorts will be tested prior to receiving drug and 90 minutes after receiving drug (midway through a three hour rest period between altitude exposures).
Time Frame: At rest, every 3 minutes during the exercise test and 5 minutes after each exercise test
Population: Not all subjects performed the same number of exercise stages to achieve VO2max.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Number analyzed (Participants) | 6 | 11 | 5
L/min
  No Drug: Rest: number analyzed (Participants) | 5 | 11 | 5
  No Drug: Rest | 8.11903 (2.05775) | 6.60219 (1.43789) | 7.53400 (1.64610)
  After Drug: Rest: number analyzed (Participants) | 5 | 9 | 4
  After Drug: Rest | 8.07571 (1.76633) | 8.98119 (2.96115) | 7.07000 (0.53110)
  No Drug: Stage 1: number analyzed (Participants) | 5 | 11 | 5
  No Drug: Stage 1 | 16.1241 (2.92554) | 14.6762 (2.51777) | 15.7480 (2.80202)
  After Drug: Stage 1: number analyzed (Participants) | 5 | 10 | 4
  After Drug: Stage 1 | 15.5680 (6.97709) | 14.7501 (2.03319) | 15.2225 (1.76415)
  No Drug: Stage 2: number analyzed (Participants) | 4 | 10 | 5
  No Drug: Stage 2 | 18.0884 (3.40527) | 16.8736 (2.56218) | 17.3880 (1.69665)
  After Drug: Stage 2: number analyzed (Participants) | 4 | 9 | 4
  After Drug: Stage 2 | 20.6211 (6.12566) | 16.8648 (2.80466) | 19.6775 (2.67616)
  No Drug: Stage 3: number analyzed (Participants) | 4 | 9 | 4
  No Drug: Stage 3 | 20.9084 (3.12626) | 18.4603 (2.61879) | 19.7900 (1.95435)
  After Drug: Stage 3: number analyzed (Participants) | 4 | 8 | 3
  After Drug: Stage 3 | 19.5537 (2.99223) | 18.0927 (3.07835) | 19.7800 (1.36173)
  No Drug: Stage 4: number analyzed (Participants) | 4 | 8 | 4
  No Drug: Stage 4 | 22.0844 (4.94934) | 20.6738 (2.60961) | 20.3775 (2.39699)
  After Drug: Stage 4: number analyzed (Participants) | 4 | 6 | 3
  After Drug: Stage 4 | 21.5792 (2.97429) | 20.8798 (1.16538) | 22.2100 (1.67189)
  No Drug: Stage 5: number analyzed (Participants) | 3 | 5 | 4
  No Drug: Stage 5 | 25.2647 (6.59397) | 22.5701 (1.61837) | 22.2475 (3.11597)
  After Drug: Stage 5: number analyzed (Participants) | 2 | 5 | 3
  After Drug: Stage 5 | 26.4806 (3.87549) | 21.9477 (1.82104) | 24.1967 (0.85008)
  No Drug: Stage 6: number analyzed (Participants) | 3 | 4 | 3
  No Drug: Stage 6 | 25.9674 (7.14490) | 22.8612 (1.49355) | 20.8800 (2.41851)
  After Drug: Stage 6: number analyzed (Participants) | 1 | 4 | 3
  After Drug: Stage 6 | 25.3863 | 23.0227 (3.22525) | 22.5067 (0.36692)
  No Drug: Stage 7: number analyzed (Participants) | 2 | 2 | 1
  No Drug: Stage 7 | 25.4212 (3.49515) | 22.0850 (2.55266) | 20.4400
  After Drug: Stage 7: number analyzed (Participants) | 0 | 2 | 0
  After Drug: Stage 7 |  | 22.5198 (5.41621) |
  No Drug: Post Exercise: number analyzed (Participants) | 3 | 10 | 5
  No Drug: Post Exercise | 10.9825 (3.61124) | 11.9949 (4.41810) | 13.9240 (4.05329)
  After Drug: Post Exercise: number analyzed (Participants) | 5 | 9 | 4
  After Drug: Post Exercise | 8.7147 (1.74727) | 10.9727 (5.02902) | 10.9875 (2.83843)

ADVERSE EVENTS:
Time Frame: 1 day or anytime after that if any complaints arose potentially attributable to the study.
Groups:
- Riociguat 0.5 mg: Riociguat 0.5 mg tablets, one-time oral dose of 0.5
  Riociguat: After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. Riociguat will be administered at the 90-minute mark of this rest period. A second VO2 max test will be repeated at altitude.
- Riociguat 1.0 mg: Riociguat 0.5 mg tablets, one-time oral dose of 1.0 mg
  Riociguat: After completion of first V02 max test at altitude, subjects will have a 3-hour rest period. Riociguat will be administered at the 90-minute mark of this rest period. A second VO2 max test will be repeated at altitude.
Arm/Group | Riociguat 0.5 mg | Riociguat 1.0 mg | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 2/11 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat 0.5 mg (N=6) | Riociguat 1.0 mg (N=11) | Control Arm (N=5)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Exercise induced
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear barotrauma (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes